CLINICAL TRIAL: NCT04836182
Title: A Double-Blind, Placebo-Controlled, Randomized, Multicenter, Phase 2 Study Assessing the Safety, Tolerability and Efficacy of IONIS-AGT-LRx, an Antisense Inhibitor of Angiotensinogen Production, Administered Subcutaneously Over 12 Weeks in Patients With Chronic Heart Failure With Reduced Ejection Fraction
Brief Title: A Study to Assess the Safety, Tolerability and Efficacy of IONIS-AGT-LRx in Participants With Chronic Heart Failure With Reduced Ejection Fraction
Acronym: ASTRAAS-HF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISIS 757456-CS5; 2020-005878-10 (EudraCT Number)
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Chronic Heart Failure With Reduced Ejection Fraction
Keywords: Heart Failure; AGT; NT-proBNP
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IONIS-AGT-LRx (Experimental): IONIS-AGT-LRX by subcutaneous injection once-weekly
  Interventions: Drug: IONIS-AGT-LRx
- Placebo (Placebo Comparator): Matching placebo by subcutaneous injection once-weekly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IONIS-AGT-LRx — Multiple doses of IONIS-AGT-LRx will be administered by SC injection.
  Other Names: ISIS 757456
  Arms: IONIS-AGT-LRx
Drug: Placebo — IONIS-AGT-LRx-matching placebo will be administered by SC injection.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of IONIS-AGT-LRX weekly subcutaneous (SC) injection on plasma angiotensinogen (AGT) concentration from Baseline to Study Day 85 (Week 13) and to evaluate the effect of IONIS-AGT-LRx weekly SC injection on plasma AGT concentration and N-terminal prohormone of B-type natriuretic peptide (NT-proBNP) levels at each scheduled visit in chronic heart failure participants with reduced ejection fraction (HFrEF).

DETAILED DESCRIPTION:
This study will be a Phase 2, double-blind, randomized, placebo-controlled study in up to 72 participants. Participants will be randomized in a 2:1 ratio to either IONIS-AGT-LRX or matching placebo and receive a once-weekly SC treatment. The length of participation in the study will be approximately 35 weeks, which includes an up to 10-week screening period, a 12-week treatment period, and a 13-week post-treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Females must be non-pregnant and non-lactating and of non- childbearing potential.
2. Males must be surgically sterile or, abstinent or, if engaged in sexual relations with a woman of child-bearing potential (WOCBP), she must be willing to use a highly effective contraceptive method
3. Screening NT-proBNP ≥ 600 picograms per milliliter (pg/mL) and less than (<) 8500 pg/mL
4. Established diagnosis of heart failure (HF) with reduced systolic function for at least 6 months prior to the screening visit (left ventricular ejection fraction, [LVEF] ≤ 40%
5. New York Heart Association class I-III

Participants should receive background standard of care for HFrEF. Therapy should have been individually optimized and stable for ≥ 4 weeks before randomization and include:

1. An angiotensin-converting-enzyme inhibitor (ACEi), or angiotensin II receptor blockers (ARBs) or sacubitril/valsartan (mandatory)
2. A beta-blocker (unless contraindicated or not tolerated)
3. A mineralocorticoid receptor antagonist (MRA, unless contraindicated or not tolerated)

Exclusion Criteria:

1. HF due to restrictive cardiomyopathy, active myocarditis, chemotherapy, hypertrophic cardiomyopathy, primary cardiac valve disease, non-compaction cardiomyopathy, or takotsubo cardiomyopathy.
2. Acute decompensated HF requiring intravenous (IV) diuretics, IV inotropes or IV vasodilators with discharge date within 30 days of screening or acute mechanical support (e.g., intra-aortic balloon pump, endotracheal intubation, mechanical ventilation, or any ventricular assist device) with discharge date within 90 days of screening.
3. Symptomatic hypotension or systolic blood pressure (SBP) ≤ 90 millimeters of mercury (mmHg) at screening.
4. Uncontrolled hypertension (HTN) (SBP > 160 mmHg or diastolic blood pressure (BP) > 100 mmHg) prior to screening.
5. Heart transplant, and/or Left Ventricular Assist Device (LVAD) prior to screening or anticipated heart transplant or LVAD during the study.
6. Implantation of a cardiac resynchronization therapy device (CRT) within 3 months prior screening or intent to implant a CRT within 3 months after screening.
7. Acute coronary syndrome, unstable angina, stroke, transient ischemic attack (TIA), coronary revascularization, cardiac device implantation, cardiac valve repair, carotid or other major surgery within 3 months of screening.
8. Coronary, valve or carotid artery disease likely to require surgical or percutaneous intervention within the 3 months after screening.
9. Severe pulmonary disease with any of the following:

   1. Requirement of continuous (home) oxygen or
   2. Known diagnosis of severe chronic obstructive pulmonary disease (as defined by the American Thoracic Society/European Respiratory Society) or severe restrictive lung disease, in the opinion of the investigator.
10. Screening laboratory results as follows, or any other clinically significant abnormalities in screening laboratory values that would render a participant unsuitable for inclusion in the opinion of the investigator.

    1. Alanine aminotransferase/aspartate aminotransferase (ALT/AST) > 2.0 × upper limit of normal (ULN).
    2. Total bilirubin ≥ 1.5 × ULN (participants with total bilirubin ≥ 1.5 × ULN may be allowed on study if indirect bilirubin only is elevated, ALT/AST is not greater than the ULN, and known to have Gilbert's disease).
    3. Platelets < 100,000/millimeter^3 (mm^3).
    4. Urine protein creatinine ratio (UPCR) ≥ 500 milligrams per gram (mg/g).
    5. Hemoglobin A1c (HbA1c) > 9.5% or uncontrolled diabetes per investigator judgement.
    6. Estimated glomerular filtration rate (eGFR) < 30 milliliters/ minute /1.73 m^2 (mL/min/1.73 meter^2) at screening.
    7. Abnormal thyroid function tests with clinical significance per investigator judgement.
    8. Serum potassium > 5.1 millimoles per liter (mmol/L) at screening.
11. Requirement of treatment with both ACEi and ARBs.
12. Previous history of intolerance to ACEi or ARBs or history of hyperkalemia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
Percent Change in Plasma AGT Concentration From Baseline to Study Day 85 | Baseline to Day 85

SECONDARY OUTCOMES:
Absolute Level of Plasma AGT | Baseline to Day 169
Change in Plasma AGT From Baseline to Each Scheduled, Post-Baseline Visit | Baseline to Day 169
Percent Change in Plasma AGT From Baseline to Each Scheduled, Post-Baseline Visit | Baseline to Day 169
Absolute Level of NT-proBNP | Baseline to Day 169
Change in NT-proBNP From Baseline to Each Scheduled, Post-Baseline Visit | Baseline to Day 169
Percent Change from Baseline in NT-proBNP to Each Scheduled, Post-Baseline Visit | Baseline to Day 169

CONTACTS AND LOCATIONS:
Locations (19):
- United States (10):
  - Arkansas Cardiology, Little Rock, Arkansas
  - Nature Coast Clinical Research - Crystal River, Crystal River, Florida
  - New Generation of Medical Research, Hialeah, Florida
  - Michigan Heart, Ypsilanti, Michigan
  - St. Louis Heart and Vascular Cardiology, St Louis, Missouri
  - The Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
  - South Oklahoma Heart Research, Oklahoma City, Oklahoma
  - Newton Clinical Research, Oklahoma City, Oklahoma
  - North Texas Research Associates, Allen, Texas
  - York Clinical Research LLC, Norfolk, Virginia
- Hungary (2):
  - Semmelweis Egyetem - Varosmajori Sziv es Ergyogyaszati Klinika, Budapest
  - Kardiologiai Maganrendeles es Klinikai Vizsgalohely, Orosháza
- Poland (7):
  - Specjalistyczna Praktyka Lekarska, Krakow
  - Samodzielny Publiczny ZOZ Centralny Szpital Kliniczny Uniwersytetu Medycznego, Lodz
  - Indywidualna Specjalistyczna Praktyka Lekarska, Lodz
  - AKA-MED Centrum Spólka z Ograniczona Odpowiedzialnoscia, Ruda Śląska
  - NZOZ Pro Cordis Sopockie Centrum Badan Kardiologicznych, Sopot
  - Centrum Chorob Serca w USK, Wroclaw
  - 4 Wojskowy Szpital Kliniczny z Poliklinika Samodzielny Publiczny ZOZ we Wroclawiu, Wroclaw

IPD SHARING:
Plan to Share IPD: No